CLINICAL TRIAL: NCT07388628
Title: ARTISTRY - ARTICE® Therapy Registry Study
Brief Title: ARTICE® Real Data Collection & Observational Trial, Phase 4 Study
Acronym: ARTistry
Status: Recruiting | Type: Observational
Sponsor: Artcline GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ARTistry
Record Dates: First submitted 2026-01-05; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sepsis; Septic Shock; Immunoparalysis in Septic Shock
Keywords: Sepsis; septic shock; Immunoparalysis in Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of this registry study are to:

1. Record real-life data related to the use of the ARTICE® therapy in sepsis subjects.
2. Further evaluate ARTICE® treatment efficacy.
3. Identify potential sub-groups, assess their risk-benefit- and safety profile.
4. Changes in SOFA score D0 to SOFA Score D7.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years who are planned to receive ARTICE® treatment during their ICU stay

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years who are planned to receive ARTICE® treatment during their ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in SOFA score D0 to SOFA Score D7 (or after last ARTICE® treatment, if later as D7). | From enrollment up to 7 days after last ARTICE® treatment.
  SOFA Score is the Sequential Organ Failure Score providing information about mortality risk, 6 organs or organ systems are assesed using specific parameters, both the sum of the points and the point development of the individual organs can be considered, normal function of organ/organ system has 0 points, severely impacted function do have 4 point, in total you can have 0 points (every organ/organ system is normale) as a minimum and 24 points as maximum (severely impacted organ/organ system)
Changes in general SOFA score and SOFA sub scores. | From enrollment up to 7 days after last ARTICE® treatment.
  SOFA Score is the Sequential Organ Failure Score providing information about mortality risk, 6 organs or organ systems are assesed using specific parameters, both the sum of the points and the point development of the individual organs can be considered, normal function of organ/organ system has 0 points, severely impacted function do have 4 point, in total you can have 0 points (every organ/organ system is normale) as a minimum and 24 points as maximum (severely impacted organ/organ system)
Changes in standard lab and inflammatory biomarkers. | From enrollment up to 7 days after last ARTICE® treatment.
  standard lab and inflammatory biomarkers for exampample are: ferritine, total bilirubin, kreatinine, CRP, lactate, gammaglobuline, amount of the different blodd cell types, like neutrophils, lymphocytes
Hospital survival rates. | From enrollment up to 7 days after last ARTICE® treatment.
Apache II Score. | From enrollment up to 7 days after last ARTICE® treatment.
  APACHE II is a clinical rating system for evaluating the severity of an illness and the risk of death in intensive care medicine; score includes information on the patient's current condition, age and concomitant diseases, values are collected over 24 hours, highest value is included in calcutaion; the score can be at minimum 0 points (lightly risk of death) and at maximum 71 (very high risk of death)
Length of ICU stay (days). | From enrollment up to 7 days after last ARTICE® treatment.
Mechanical ventilation days. | From enrollment up to 7 days after last ARTICE® treatment.
Renal replacement therapy days. | From enrollment up to 7 days after last ARTICE® treatment.
Vasopressor therapy days. | From enrollment up to 7 days after last ARTICE® treatment.
Frequency of secondary infections. | From enrollment up to 7 days after last ARTICE® treatment.
Type of secondary infections: it will be divided into viral, bacterial or fungi infection. | From enrollment up to 7 days after last ARTICE® treatment.
  It is recorded whether the infection is viral, bacterial, or caused by fungi. And in case of bacterial infection it will be recorded weather, it is gram-positive or gram-negative bacterial infection.
Changes in the physiological parameter heartrate. | From enrollment up to 7 days after last ARTICE® treatment.
  as physiological parameter will be measured heartrate in bpm
Changes in physiological parameter blood pressure. | From enrollment up to 7 days after last ARTICE® treatment.
  as physiological parameter will be measured systolic and diastolic blood pressure in mmHg.
Changes in physiological parameter body temperature. | From enrollment up to 7 days after last ARTICE® treatment.
  as physiological parameter will be measured body temperature in °C
Changes in physiological parameter mean arterial pressure. | From enrollment up to 7 days after last ARTICE® treatment.
  as physiological parameter will be measured mean arterial pressure in mmHG
Complications related to the ARTICE® therapy application. | From enrollment up to 7 days after last ARTICE® treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sauer, Prof. Dr. med., Principal Investigator — Klinikum Magdeburg, Klinik für Intensiv- & Rettungsmedizin
Locations (1):
- Klinikum Magdeburg, Klinik für Intensiv- und Rettungsmedizin, Magdeburg, Germany